CLINICAL TRIAL: NCT00058760
Title: A Randomized Controlled Trial of the NIA Intervention
Brief Title: Delaying Sexual Activity in African American Adolescent Girls
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HD39757-1; 1R01HD039757 (NIH)
Record Dates: First submitted 2003-04-11; First posted 2003-04-15 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-03

CONDITIONS: Adolescent Behavior; Sex Behavior
Keywords: Prevention of early sexual behavior; NIA intervention
MeSH Terms: conditions — Adolescent Behavior; Sexual Behavior

INTERVENTIONS:
Behavioral: NIA intervention (after school health promotion didactic program)

SUMMARY:
This study will evaluate the effectiveness of a program designed to prevent early sexual behavior in middle school-aged African American girls.

DETAILED DESCRIPTION:
There are 34 million adolescents between the ages of 11 and 17 years old in the United States. Approximately 12% of them are African American. These youths experience earlier pubertal onset and face earlier challenges to participate in sexual activity, and therefore have earlier potential for pregnancy and contraction of sexually transmitted diseases. Experts in adolescent research have recommended developing and implementing new interventions to reduce early sexual activity; these interventions should target middle school-aged youths. The purpose of this study is to evaluate the efficacy of the NIA intervention on intention to engage in early sexual behavior and actual involvement in early sexual behavior in a convenience sample of sixth and seventh grade African American girls.

NIA is a Swahili word that means "having a sense of purpose." It is one of the seven principles of Kwanzaa, a holiday that celebrates African Americans' cultural roots in Africa. The intervention was named after a self-development program for African American girls to highlight the intervention's cultural basis.

The study will provide 12 weekly and 5 booster after school didactic sessions; these sessions will teach health promotion and decision making skills to help girls successfully avoid situations where sexual activity is invited. Mothers and daughters will collaborate on homework assignments on puberty, heterosexual relationships, and sexual issues. The study will provide an evening mother-daughter workshop on sexual responsibility and a "Baby-Think-It-Over" weekend experience for girls using a computerized doll. Finally, the study will provide five "Hey Baby!" role-play vignettes to teach girls how to avoid heterosexual relationships that may lead to sexual activity.

The NIA intervention will be compared against a usual after-school activity control group of sixth and seventh grade African American girls in two public middle schools in the Pittsburgh Public School system. Participants will be randomly assigned to either the NIA intervention group or the control group. Each participant will be in the study for 1 year. There will be a 12-week main intervention in the fall, a 5-week booster in the spring, and final testing 1 year after study entry. Assessments will be primarily paper and pencil tests of the study's main outcome variables: attitude toward early sexual behavior (ESB); subjective norms (mother, father, peer) toward ESB; intention to engage in ESB; and self-reported ESB. Additionally, there will be knowledge content quizzes after each main intervention or booster session and a written evaluation of the "Baby-Think-It-Over" weekend.

ELIGIBILITY:
Inclusion Criteria

* African American
* 11 to 14.3 years old

Exclusion Criteria

* Participation in similar programs, such as Best Friends or Postponing Sexual Involvement
* Classification in school as a special education student
* Anorexia, bulimia, or chronic or acute reproductive health disease
* Prior or current pregnancy
* Prior participation in the community NIA girls' program

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240
Dates: Start 2001-02; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Willa Doswell, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Dr. Willa Doswell, Pittsburgh, Pennsylvania, United States